CLINICAL TRIAL: NCT05715645
Title: Assessment of Recovery After Adductor Canal Block Analgesia Associated Either With Infiltration Between Popliteal Artery and Posterior Capsule, or With Surgical Peri-articular Infiltration for Patients Treated by Improved Recovery Program
Brief Title: Assessment of Recovery After Adductor Canal Block Analgesia in Unilateral Prosthetic Knee Surgery
Acronym: IPACKNEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022-A01884-39
Record Dates: First submitted 2023-01-26; First posted 2023-02-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Unilateral Primary Osteoarthritis of Knee
MeSH Terms: interventions — Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient and the people carrying out the functional assessments (physiotherapists) will be blinded to the analgesia received, unlike the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block at the Adductor Canal + Infiltration between Popliteal Artery and Posterior Capsule (Experimental): Adductor canal block analgesia associated with infiltration between the popliteal artery and the posterior capsule
  Interventions: Procedure: Unilateral prosthetic knee surgery; Procedure: Analgesia
- Block at the Adductor Canal + High Volume Local Infiltration Analgesia (Active Comparator): Adductor canal block analgesia associated with surgical periarticular infiltration
  Interventions: Procedure: Unilateral prosthetic knee surgery; Procedure: Analgesia

INTERVENTIONS:
Procedure: Unilateral prosthetic knee surgery — Unilateral prosthetic knee surgery
Procedure: Analgesia — Analgesic management by adductor canal block

SUMMARY:
The purpose of the study is post-operative recovery from prosthetic knee surgery will be assessed by the proportion of patients entering the Accelerated Rehabilitation After Surgery program eligible for discharge from hospital at 2 days according to the following definition: Chung score ≥ 9 with no intravenous (IV) infusion, solid food, transit restored, no signs of infection and Cumulated Ambulation Score D1 ≥ 5 (if discharged on Day 1), Cumulated Ambulation Score Day 2 ≥ 10 (if discharged on Day 2), or Cumulated Ambulation Score Day 3 ≥ 11/18.

DETAILED DESCRIPTION:
This is a monocentric, interventional, prospective, comparative, randomized study in 2 parallel groups, single-blind. The study is proposed to the patient during the preoperative anesthetic consultation. The patient and the people carrying out the functional assessments (physiotherapists) will be blinded to the analgesia received, unlike the investigator.

Patients will be included by an anesthesiologist during the preoperative anesthetic consultation. After the Accelerated Rehabilitation After Surgery consultation, they will then be operated on (Day 0) and seen up to 5 times post-operatively over a period of 45 days for the purposes of the study: at 24h, 48h, 72h, discharge from hospital and 45 days post operative. Discharge from hospital occurs during follow-up depending on the patient's condition. These visits will coincide with follow-up consultations with the surgeon as part of the usual management.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a score "American Society of Anesthesiologists" I to III;
* Patient undergoing initial unilateral prosthetic knee replacement surgery for osteoarthritis;
* Patient eligible for analgesia by block of the adductor canal associated with additional infiltration;
* Patient accepting to follow the enhanced recovery program after surgery;
* Patient who signed an informed consent form to participate in the study.

Exclusion Criteria:

* Patient with a known allergy to a study product;
* Patient having undergone previous surgery with a prosthesis on the knee to be operated on;
* Patient with morbid obesity (Body Mass Index > 40);
* Patient with a pre-existing inability to walk;
* Patient with a history of chronic neuropathic pain in the leg undergoing surgery;
* Patient with heart failure with impaired ejection fraction;
* Patient with a history of drug addiction;
* Patient chronically taking level III analgesics;
* Patient taking gabapentin or pregabalin chronically;
* Patient with severe renal or hepatic impairment;
* Patient with a high level of dependence, defined by level 1 or 2 of the Iso-Ressources Group;
* Protected patient (under legal protection, or deprived of liberty by judicial or administrative decision);
* Patient unable to understand the information related to the study (linguistic, psychological, cognitive reasons, etc.);
* Pregnant or likely to be pregnant (of childbearing age without effective contraception) or breastfeeding;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient not benefiting from a social security scheme.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative recovery from knee prosthesis surgery | 3 days
  Post-operative recovery from prosthetic knee surgery will be assessed by the proportion of patients entering the Accelerated Rehabilitation After Surgery program eligible for discharge from hospital at 2 days according to the following definition: Chung score ≥ 9 with no intravenous (IV) infusion, solid food, transit restored, no signs of infection and Cumulated Ambulation Score D1 ≥ 5 (if discharged on Day 1), Cumulated Ambulation Score Day 2 ≥ 10 (if discharged on Day 2), or Cumulated Ambulation Score Day 3 ≥ 11/18.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Médipôle, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No